CLINICAL TRIAL: NCT05982925
Title: Longitudinal Investigation of Cortical Demyelination and Meningeal Inflammation in Multiple Sclerosis and Related Disorders
Brief Title: Longitudinal Cortical Demyelination in Multiple Sclerosis and Related Disorders
Status: Enrolling by invitation | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Erin Beck, Assistant Professor of Neurology, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-21-01855
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis; Neuromyelitis Optica; Demyelinating Autoimmune Diseases, CNS
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica; Demyelinating Autoimmune Diseases, CNS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- MS Participant: Adults with multiple sclerosis
- Control Participant: Adults without neurologic disease
- Other Neuroinflammatory Participants: Adults with a neuroinflammatory disease that is not multiple sclerosis

SUMMARY:
In this protocol, a combination of MRI, blood, and cerebrospinal fluid (CSF) analysis will be used to understand the natural history, underlying immunologic mechanisms, and clinical implications of central nervous system (CNS) lesions, in particular lesions in the cerebral cortex, in multiple sclerosis (MS) and other inflammatory and autoimmune disorders affecting the CNS. Patients with these disorders, as well as healthy controls, will undergo baseline clinical evaluation and testing, bloodwork, and MRI, with follow up clinical evaluation, bloodwork, and MRI at years 1, 3, and 6. Additional MRIs may be performed in patients with possible new lesion formation or to compare MRI techniques. Lumbar puncture will be performed on participants who are not currently being treated with disease modifying therapies and who are willing to undergo the procedure.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* able to provide consent in English
* able to undergo MRI

Exclusion Criteria:

* contraindication to MRI
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with MS or other neuroinflammatory diseases and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2034-07-31 (Estimated)

PRIMARY OUTCOMES:
Cortical Lesion Number | at 6 years (end of study)
  Lesions in the cerebral cortex

CONTACTS AND LOCATIONS:
Overall Officials: Erin S Beck, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. Any purpose. Specify Other Mechanism Proposals should be directed to erin.beck@mssm.edu To gain access, data requestors will need to sign a data access agreement.